CLINICAL TRIAL: NCT01477255
Title: The Feasibility Of a Daily Diary Methodology With a Pediatric Cancer Population: A Pilot Study
Brief Title: The Feasibility Of a Daily Diary Methodology With a Pediatric Cancer Population
Acronym: DIARY1
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DIARY1
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: daily assessment; electronic diary; coping strategies; resiliency of cancer patients; psychology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cancer patient: Patient participants will include children and adolescents between the ages of 8-17 years who have been recently diagnosed with cancer. They will use an iPad as a diary to track their daily experiences. They will use an iPad as a diary to track their daily experiences.
  Interventions: Behavioral: iPad
- Control: For each pediatric patient enrolled, a child without a history of a serious medical illness will be recruited from the larger community who is matched on variables of age, race/ethnicity, gender, and socioeconomic status. They will use an iPad as a diary to track their daily experiences. They will use an iPad as a diary to track their daily experiences.
  Interventions: Behavioral: iPad

INTERVENTIONS:
Behavioral: iPad — The proposed investigation is a prospective case-control pilot study. The major goal of this pilot study is to assess the feasibility of a daily diary methodology for monitoring the experiences of recently diagnosed pediatric cancer patients and healthy-matched peers. The investigation will also examine the relationships among individual and contextual factors that influence the daily psychosocial functioning of youth with cancer in comparison to youth without cancer.
  Other Names: electronic diary

SUMMARY:
This investigation seeks to determine the feasibility of an electronic diary methodology among pediatric cancer patients and healthy matched controls. Levels of study participation and compliance will be assessed to assist with determining overall feasibility. Results will offer insight into the effectiveness of this means of data collection with a pediatric oncology population, and will examine how psychosocial and contextual factors contribute to the resiliency that has been demonstrated by children with cancer. Findings will provide data for the design and implementation of a future, larger-scale study with this pediatric population that implements an electronic daily diary methodology.

DETAILED DESCRIPTION:
The study will include two phases of participant recruitment and participation. Phase I will include recruitment of six pediatric patients to pilot an electronic daily diary on an Apple iPad. These participants will be prompted by the iPad once daily for seven days, and will be asked to answer multiple choice and yes/no questions related to their daily experiences, activities and emotions. Following the week of daily diary completion, each participant in Phase I will engage in a brief feedback interview with a member of the research team to discuss his/her overall experiences using the electronic diary, including any technological issues that arise. The purpose of Phase I is to work out any technological and/or logistical problems associated with completion of the daily iPad diary.

After any technological problems have been addressed, Phase II of the study will begin. Child participants in Phase II of the study will complete several paper and pencil questionnaires on two separate occasions that assess factors including optimism, experience of various emotions, spirituality, relationships with others, benefit-finding, quality of life, and resiliency. Children will also complete two weeks of daily electronic diaries that will prompt them to answer multiple choice and yes/no questions related to their daily experiences, activities and emotions. One parent or guardian will also be recruited to participate, and will complete paper and pencil questionnaires on two separate occasions that ask about optimism, the parent-child relationship, spirituality, psychological functioning, and their perceptions of their children's behavior and mood.

Finally, following the completion of the first week of daily diaries, a short interview will be conducted with each child and parent dyad to gather information about the child's experiences using the electronic diary. They will be asked to provide feedback about any challenges and technological difficulties that they encountered, as well as their general thoughts about using the electronic diary. The interview will also include an opportunity to trouble-shoot difficulties associated with using the electronic daily diary in preparation for the second week of diary completion. For each participant, we anticipate a participation timeframe of 10-15 weeks.

Primary Objective:

* To evaluate the usefulness of an electronic daily diary for understanding the experiences, emotions, and coping strategies of children with cancer and of their healthy peers.

ELIGIBILITY:
Inclusion Criteria for Pediatric Participants:

* Research participant is between ages 8 and 17 years inclusive.
* Research participant has received a diagnosis of malignancy in the period 10 weeks prior to enrollment.
* Research participant has no significant cognitive, motor, or sensory deficits that would preclude completion of the study measures.
* Research participant is able to speak and read English.

Inclusion Criteria for Control Participants:

* Research participant is between ages 8 and 17 years inclusive.
* Research participant has no history of a major medical diagnosis.
* Research participant has no significant cognitive, motor, or sensory deficits that would preclude completion of the study measures.
* Research participant is able to speak and read English.

Exclusion Criteria:

* Participants are excluded if they fail to meet any of the Inclusion Criteria for Pediatric or Control Participants.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All eligible participants will be invited to participate in the research investigation, including children and parents of both genders and of all races/ethnicities.
  St. Jude treats pediatric patients from across the country and around the world, which results in a culturally diverse pediatric population. Based upon enrollment patterns from previous investigations, it is anticipated that approximately 19% of enrolled pediatric participants will be racial/ethnic minority children. Because the control group will be matched to the pediatric group on variables of gender, age, race/ethnicity, and socioeconomic status, it is anticipated that the gender and race/ethnicity of the control group will be commensurate with that of the pediatric group.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2011-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The number who agree to participate compared to the total number approached for the study. | Day 0 of study
  The rate of agreement to participate in the study.
The number of total days the participant was able to complete the daily diary. | From on-study date through up to 4 months
  The rate of completion of daily diary measures, and the number of participants who complete the study in its entirety.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Phipps, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols